CLINICAL TRIAL: NCT07389070
Title: Evaluating the Effectiveness of Positional Release Technique With and Without Therapeutic Exercises for Chronic Low Back Pain Management
Brief Title: Positional Release With/Without Exercise for Chronic LBP
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palestine Ahliya University (Other)
Responsible Party: Principal Investigator, Azzam Alarab, Azzam M. Alarab, Ph.D Assistant Professor Chairperson, Department of Medical Sciences - Master's Palestine Ahliya University, Palestine Ahliya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAU
Record Dates: First submitted 2026-01-24; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Back Disorder
Keywords: LBP; PRT; Exercies
MeSH Terms: interventions — Hypoxanthine Phosphoribosyltransferase; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1- Group A (PRT): Positional Release Technique with exercises (Experimental): Group A (n=30) underwent a 12-session program over four weeks. Each 40-minute session combined two 30-minute positional release procedures with three 10-minute therapeutic exercise modules.
  Interventions: Other: PRT with exercises
- arm 2- Group A (PRT): Positional Release Technique without exercises (Experimental): Group B received 12 treatment sessions over four weeks (three sessions/week), each consisting of two positional release procedures totaling 30 minutes.
  Interventions: Other: PRT Without exercises

INTERVENTIONS:
Other: PRT with exercises — Postional release technique with exercises.
  Arms: arm 1- Group A (PRT): Positional Release Technique with exercises
Other: PRT Without exercises — Postional release technique without exercises.
  Arms: arm 2- Group A (PRT): Positional Release Technique without exercises

SUMMARY:
Chronic low back pain (CLBP) presents a significant therapeutic challenge due to its multifactorial nature and high recurrence rate. While manual therapy techniques like Positional Release Technique (PRT) are commonly employed to modulate pain and improve tissue function, there is a growing consensus in rehabilitation that their effects may be transient if not coupled with active strategies to address underlying impairments. Therapeutic exercises (TE) form a cornerstone of CLBP management by aiming to restore strength, endurance, and neuromuscular control. However, the specific additive benefit of combining a passive, indirect technique like PRT with a structured TE program remains an area for empirical investigation. This study, therefore, sought to compare the clinical effectiveness of an integrated approach using PRT alongside TE against the application of PRT alone, hypothesizing that the combined intervention. would yield superior outcomes in pain reduction and functional improvement for individuals with CLBP.

DETAILED DESCRIPTION:
Background & Rationale:

Chronic low back pain (CLBP) is complex and prone to recurrence, making its management difficult. Clinicians often use passive manual therapies like the Positional Release Technique (PRT) to reduce pain. However, evidence suggests that passive treatments alone may not provide long-term relief unless combined with active interventions. Therapeutic exercise (TE) is a fundamental active approach that targets core deficits in strength and motor control. The key question is whether adding TE to PRT offers a significant advantage over PRT used in isolation.

Aim:

This study aimed to directly compare the clinical effectiveness of a combined treatment (PRT + TE) versus PRT alone in managing CLBP, with the hypothesis that the combined approach would be superior.

Methodology:

A randomized controlled trial was conducted with 60 participants diagnosed with CLBP (pain duration ≥3 months), aged 20-65. They were recruited from a single physiotherapy center. Participants with specific spinal pathologies (e.g., fractures, disc abnormalities) were excluded. They were randomly divided into two groups:

Group A (Experimental): Received PRT combined with a structured Therapeutic Exercise program.

Group B (Control): Received PRT alone.

Outcome Measures:

Effectiveness was assessed using standardized tools measured before and after the treatment period:

Pain Intensity: Visual Analogue Scale (VAS). Functional Disability: Roland-Morris Questionnaire (RMQ). Muscular Performance: A curl-up test for abdominal endurance.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 20-65 years.
* Clinical diagnosis of chronic low back pain (CLBP).
* Positive Faber (Patrick's) test.
* Positive Slump test.
* A pain intensity score of ≥3 on the Visual Analogue Scale (VAS).
* Symptoms presenting with or without referred leg pain.

Exclusion Criteria:

* Diagnosis of spondylolisthesis, disc disease, osteoporosis, or other significant bone disease.
* History of vertebral fractures.
* History of spinal surgery.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
VAS | 4 weeks
  A validated, single-item scale used to measure subjective pain intensity. Patients mark a point on a 10-cm line anchored by "no pain" (0) and "worst pain imaginable" (10). The score is the measured distance in cm/mm, providing a quantitative pain rating.
RMQ | 4 weeks
  The Roland-Morris Disability Questionnaire (RMQ) is a widely used, self-administered, health status measure designed to assess physical function and disability specifically related to low back pain. It consists of 24 yes/no statements derived from the Sickness Impact Profile, each describing a specific activity limitation due to back pain (e.g., "I walk more slowly because of my back"). The total score (0-24) is the sum of items marked "yes," with a higher score indicating greater disability. It is valued for its brevity, ease of use, and responsiveness to clinical change.
Endurance | 4 weeks
  An endurance test is a performance-based assessment that measures the ability of specific muscle groups (particularly the trunk stabilizers: back extensors, flexors, and lateral musculature) to maintain a submaximal contraction or a fixed posture against gravity over time. Common examples used in low back pain research include the prone plank (trunk flexors), Sorensen/Biering-Sørensen test (back extensors), and side plank (lateral stabilizers). The outcome is the time (in seconds) the position can be held until failure, providing an objective measure of muscular stamina.

CONTACTS AND LOCATIONS:
Locations (1):
- Palestine Ahliya University, Bethlehem, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] https://doi.org/10.1056/NEJMcp2032396